CLINICAL TRIAL: NCT06136286
Title: Effects of Blood Flow Restriction Rehabilitation After ORIF of Distal Radius Fractures
Brief Title: ORIF Distal Radius Blood Flow Restriction Therapy
Acronym: ORIF DR BFR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shari Liberman, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro000022755
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: The study will be a prospective randomized control trial consisting of subjects requiring ORIF of the distal radius. Subjects will be divided into two groups based on age, then subsequently be randomly divided into two groups following their inclusion in the study. Group 1) Control group in which subjects receive standard of care rehab. Group 2) BFR group in which BFR is incorporated into the patients' rehab.
  Groups will be normalized based on gender. One group will undergo the normal rehabilitation protocol for the hand and wrist as determined by Dr. Liberman. The study group will undergo rehabilitation protocol for distal radius fractures modified by use of a tourniquet for blood flow restriction during selected exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): Standard of care postoperative rehabilitation. Subject will undergo standard rehab following surgery without BFR.
- Intervention - Blood Flow Restriction Therapy (BFR) (Experimental): Subjects will undergo standard postoperative rehabilitation that incorporates BFR during certain exercises.
  Interventions: Device: Blood Flow Restriction (BFR) Cuff

INTERVENTIONS:
Device: Blood Flow Restriction (BFR) Cuff — The intervention group will receive therapy with a blood flow restriction cuff that restricts blood flow at their individual limb occlusion pressure during specific exercises.
  Arms: Intervention - Blood Flow Restriction Therapy (BFR)

SUMMARY:
Patients commonly experience a significant amount of muscular atrophy following open reduction internal fixation (ORIF) surgery of distal radius fractures, associated with an increased risk of re-injury, and an increase in time of recovery. A combination of low intensity resistance exercise and blood flow restriction (BFR) therapy has been shown to elicit responses similar to high intensity resistance exercise with reduced risk. We hypothesize that chronic low intensity resistance exercise combined with BFR will improve muscular strength, reduce skeletal muscle atrophy, and will enhance recovery.

Therefore, the specific aims of this study are as follows:

1. Determine if BFR added to standard post-operative rehab will prevent skeletal muscle atrophy and promote skeletal muscle growth during 12-weeks of rehab training compared to traditional rehab alone. The working hypothesis, founded on previous literature, is that combined rehab and BFR will enhance skeletal muscle growth and prevent atrophy to a greater extent than rehab alone.
2. Determine if BFR added to standard post-operative rehab will improve muscular strength following surgery compared to traditional rehab alone. Because strength can be attributed to skeletal muscle mass, the working hypothesis, founded on previous literature, is that combined rehab and BFR will enhance skeletal muscle strength and fatigue resistance to a greater extent than rehab alone.
3. Determine if BFR added to standard post-operative rehab will improve functional outcomes following surgery compared to traditional rehab alone. The working hypothesis, founded on previous literature is that BFR will improve functional outcomes over rehab alone.

DETAILED DESCRIPTION:
he study will be a prospective randomized control trial consisting of subjects requiring ORIF of the distal radius. Subjects will be divided into two groups based on age, then subsequently be randomly divided into two groups following their inclusion in the study.

Groups will be normalized based on gender. One group will undergo the normal rehabilitation protocol for the hand and wrist as determined by Dr. Liberman. The study group will undergo rehabilitation protocol for distal radius fractures modified by use of a tourniquet for blood flow restriction during selected exercises. On the day of the procedure, the surgeon will measure the subject's forearm girth, the location of the largest circumference. The subject will then undergo the normal operative fixation of the distal radius fracture. A subject will be excluded from the study if they have had any prior surgeries on their affected wrist. At the subject's two week postoperative clinic visit, the physician will measure forearm girth. Study group subjects will begin physical therapy instructed BFR exercises at two weeks post operatively. Study group subjects will be taken through normal hand and wrist rehab protocol as well as BFR exercises. Control group subjects will do the same exercises and formal physical therapy rehab protocol as the study group without BFR.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18+
* With acute fracture of distal radius requiring ORIF surgery

Exclusion Criteria:

* Exorbitant pain (VAS >8/10) related or unrelated to exercise
* Prior trauma or surgery to the observed limb
* Level 2 Obesity (BMI>35)
* Diabetes - Type II
* Cardiovascular, renal, liver or pulmonary disease
* Active infections
* Cancer (current or treated within the past 2 years)
* Bleeding or coagulation disorder
* Rapid weight change within the past year
* Physically unable to participate in the intervention
* Currently taking, or recently (w/in 1month of participation) taken prescribed or over the counter ergogenic aids or compounds known to be banned by the NCAA
* Unable to complete a minimum of 85% of the assigned rehabilitation sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Body composition / bone density | DEXA scans will be recorded at the first rehabilitation visit (one week post-op), and then at two weeks, six weeks and 12 weeks following the initiation of rehabilitation.
  Soft tissue analysis of forearm and total body via DEXA scan.
Forearm girth | Measurements will be recorded on the day of operative procedure, then at two, six and 12 weeks post-op.
  The location of the largest circumference will be measured by the operating surgeon. Values recorded in cm.
Grip strength | Measurements will be recorded on the day of operative procedure, then at two, six and 12 weeks post-op.
  Grip strength will be measured for both left and right hands using a handheld dynamometer. Values recorded in lbs.
Pinch grip strength | Measurements will be recorded on the day of operative procedure, then at two, six and 12 weeks post-op.
  Pinch grip strength will be measured for both left and right hands using a handheld dynamometer. Values recorded in lbs.

SECONDARY OUTCOMES:
DASH survey | This survey will be conducted before surgery, prior to physical therapy rehabilitation at two weeks post-op, then at two months, six months and one year post-operatively.
  Patient reported outcome surveys will be completed by all participants to measure information relating to pain/symptoms and functional ability post-op.
Michigan Hand Outcomes survey | This survey will be conducted before surgery, prior to physical therapy rehabilitation at two weeks post-op, then at two months, six months and one year post-operatively.
  Patient reported outcome surveys will be completed by all participants to measure information relating to pain/symptoms and functional ability post-op.
Patient Rated Wrist Evaluation | This survey will be conducted before surgery, prior to physical therapy rehabilitation at two weeks post-op, then at two months, six months and one year post-operatively.
  Patient reported outcome surveys will be completed by all participants to measure information relating to pain/symptoms and functional ability post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Liberman, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No